CLINICAL TRIAL: NCT02024165
Title: Electrode-Based Sensor for Non-Invasive Fetal Heart Rate Monitoring With Improved Reliability
Acronym: FHR
Status: Completed | Type: Observational
Sponsor: OBMedical Company (Other)
Responsible Party: Sponsor
Other Study IDs: OBM-WP-2013; IRB (Other: 510126-1)
Record Dates: First submitted 2013-12-02; First posted 2013-12-31 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-04

CONDITIONS: Laboring Women With Ultrasound and FSE Monitoring
Keywords: Ultrasound; FSE; IUPC

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Electrode Sensor, FSE: Pregnant women between the ages of 18-50 with a single viable fetus in cephalic presentation monitored with Electrode Sensor, and/or FSE
- Electrode Sensor, Ultrasound: Pregnant women between the ages of 18-50 with a single viable fetus in cephalic presentation monitored with Electrode Sensor, and/or Ultrasound

SUMMARY:
The specific goal of the proposed research is to develop a reliable, non-invasive fetal and maternal heart rate and contraction monitor that is unaffected by obesity and requires less nursing intervention than the tocodynamometer and Doppler ultrasound.

DETAILED DESCRIPTION:
The majority of obstetric deliveries in the US undergo electronic monitoring and continuous uterine activity and fetal heart rate (FHR) monitoring is the standard of care. Typically, external transducers are employed, the reliability of which depends on their proper positioning, which may be disturbed by patient or fetal movement. The tocodynamometer (strain gauge, toco for short) provides frequency and timing of contractions, but requires transmission of tension from the uterus to the sensor. Fetal heart rate is acquired with an external Doppler ultrasound transducer. The reliability of this monitor depends on the ability to obtain a window to the fetal heart.

In some patients, particularly the obese, the toco and ultrasound may fail to monitor consistently. In others both transducers require frequent repositioning by the nursing staff, and the Doppler may erroneously report maternal heart rate instead of fetal.

The alternative uterine activity monitor is an intrauterine pressure catheter (IUPC), which is placed through the cervical os in the adequately dilated patient with ruptured membranes. While this monitor usually provides a more reliable signal than the toco, as well as quantitative information regarding intrauterine pressure, it is invasive and there is an increased risk of infection. The alternative FHR monitor is via fetal scalp electrode (FSE), which is applied transvaginally to the fetal presenting part, also requiring adequate cervical dilation and ruptured membranes. While the FSE usually provides a more reliable signal, it is similarly invasive and increases risk of infection.

Maternal obesity (defined as BMI at presentation ≥ 30) is an ever-increasing problem in the US, and is even more prominent in the obstetric suite. Meanwhile, obese women have an increased risk for labor problems, infections and other complications. Noninvasive labor monitoring, while preferable to reduce the infection risk, is particularly unreliable in this population.

ELIGIBILITY:
Inclusion Criteria:

* Parturients presenting to Labor & Delivery for labor at term (>36 weeks completed gestation)
* Single viable fetus in cephalic presentation
* With FSE or IUPC for obstetric indications

Exclusion Criteria:

* Multi fetal gestation
* Contraindication to FSE or IUPC placement
* Insufficient abdominal space for all required sensors

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Laboring women in Labor and Delivery Ward
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Busowski, MD, Principal Investigator — Winnie Palmer Hospital for Women and Babies
Locations (1):
- Winnie Palmer Hospital for Women and Babies, Orlando, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Electrode Sensor, FSE, Ultrasound: Pregnant women between the ages of 18-50 with a single viable fetus in cephalic presentation monitored with Electrode Sensor, and/or FSE and Ultrasound
Period: Overall Study
Arm/Group | Electrode Sensor, FSE, Ultrasound
Started | 71
Completed | 71
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Electrode Sensor, FSE, Ultrasound: Pregnant women between the ages of 18-50 with a single viable fetus in cephalic presentation monitored with Electrode Sensor and/or FSE and Ultrasound
Arm/Group | Electrode Sensor, FSE, Ultrasound
Number analyzed (Participants) | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 71
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 71

OUTCOME MEASURES:

1. Primary Outcome: Fetal Heart Rate Interpretability
Description: The Fetal Heart Rate (or FHR) of the electrode sensor will be compared to the FHR of the ultrasound when both are compared to the FSE. Percentage of time that signals are interpretable will be compared between devices
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: percentage of time the signals are inter
Arm/Group | Electrode Sensor, FSE | Electrode Sensor, Ultrasound
Number analyzed (Participants) | 71 | 71
percentage of time the signals are inter | 83.4 (15.4) | 62.4 (26.7)

ADVERSE EVENTS:
Arm/Group | Electrode Sensor, FSE, Ultrasound
Serious Adverse Events (participants affected / at risk) | 0/71
Other Adverse Events (participants affected / at risk) | 0/71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No